CLINICAL TRIAL: NCT01930682
Title: EARLY Routine Catheterization or Rescue Angioplasty After Alteplase Fibrinolysis vs. Primary Angioplasty in Acute ST-elevation MYOcardial Infarction: An Open, Prospective, Randomized, Multicentre Trial
Brief Title: EARLY Routine Catheterization After Alteplase Fibrinolysis vs. PPCI in ST-Segment-Elevation MYOcardial Infarction
Acronym: EARLY-MYO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BI135.326; 12410708300 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2013-08-19; First posted 2013-08-29 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2013-08

CONDITIONS: Acute ST-segment Elevation Myocardial Infarction
Keywords: Myocardial Infarction; Catheterization; Fibrinolysis
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early post-fibrinolytic catheterisation (Experimental): For STEMI Patients, alteplase is given as a intravenous bolus (8-mg) followed by 42 mg iv gtt in 90 min.Early routine catheterization after 3 hours but within 24 hours of the start of fibrinolytic therapy is performed, if required, PCI or, in case of insufficient ST resolution at 90 min,rescue PCI. The decision on rescue PCI will, however, be taken 90 min (or earlier if clinically indicated) after injection of alteplase according to the ST resolution (less than 50% reduction in ST-segment elevation).
  Interventions: Drug: Alteplase; Procedure: Early post-fibrinolytic catheterisation
- Primary PCI (Other): For STEMI Patients,primary PCI is performed without fibrinolytic therapy.
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Drug: Alteplase — Alteplase is given as a intravenous bolus (8-mg) followed by 42 mg iv gtt in 90 min.
  Other Names: rt-PA
  Arms: Early post-fibrinolytic catheterisation
Procedure: Early post-fibrinolytic catheterisation — Early post-fibrinolytic catheterisation after 3 hours but within 24 hours of the start of fibrinolytic therapy is performed, if required, PCI or, in case of insufficient ST resolution at 90 min,rescue PCI. The decision on rescue PCI will, however, be taken 90 min (or earlier if clinically indicated) after injection of alteplase according to the ST resolution (less than 50% reduction in ST-segment elevation).
  Arms: Early post-fibrinolytic catheterisation
Procedure: Primary PCI — For STEMI Patients,primary PCI is performed within 12 hours after the onset.
  Arms: Primary PCI

SUMMARY:
The EARLY-MYO (EARLY routine catheterization after alteplase fibrinolysis vs. primary PCI in acute ST-segment elevation MYOcardial infarction) is an investigator-initiated, prospective, multicenter, randomized (1:1), open-label, actively-controlled, parallel group, non-inferiority trial comparing the efficacy and safety of a PhI strategy with half-dose fibrinolysis versus PPCI in STEMI patients presenting within 6 hours after symptom onset and with an expected PCI-related delay of ≥60 min.

DETAILED DESCRIPTION:
Early, successful restoration of myocardial perfusion after a ST-elevation myocardial infarction (STEMI) is the most effective way to reduce final infarct size and improve clinical outcome. Reperfusion for STEMI treatment in the modern era encompasses mechanical and pharmacological strategies. It is generally well-accepted that primary percutaneous coronary intervention (PPCI) is the preferred reperfusion strategy for all STEMI patients when it can be performed within the guideline-recommended timeframe at PPCI-capable facilities. However, PPCI is not universally available, and delays in performing percutaneous coronary intervention (PCI) are common in real-world practice. Even in some large cities, patients have a high chance of presenting to hospitals not providing around-the-clock PPCI service. Given this background, in recent years there has been great interest and progress in creating triage strategies for STEMI patients who cannot receive timely PPCI.

Pharmaco-invasive (PhI) strategy, an early reperfusion strategy by initial prompt fibrinolysis with subsequent early catheterization (with either routine early PCI after successful fibrinolysis or rescue PCI as needed), has been proposed as a therapeutic option for STEMI patients when timely PPCI is not feasible. However, current evidence on the efficacy and safety of PhI strategy in STEMI patients is limited, and the role of PhI strategy in STEMI continues to be debated. Given that no randomized clinical trial is available to compare a PhI strategy with half-dose fibrinolytic regimen versus PPCI in STEMI patients, investigators plan to perform a controlled, randomized trial to evaluate the efficacy and safety of a PhI strategy with half-dose alteplase fibrinolysis versus PPCI in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 or 18 years old, less than 75 years old;
* Patents with myocardial infarction who have symptom onset within 6h before randomization;
* ECG: ≥2 mm ST-segment elevation in 2 contiguous precordial leads or ≥1 mm ST-segment elevation in 2 contiguous extremity leads ;
* Patents with an expected PCI-related delay [expected time delay from FMC to first balloon dilation≥90 min, and difference between the time of FMC to balloon dilation minus the time from FMC to start of fibrinolysis ≥60 minutes)];
* Signed informed consent form prior to trial participation.

Exclusion Criteria:

1. Evidence of cardiac rupture;
2. ECG: new left bundle branch block;
3. "Diagnosis to balloon inflation" time over 3 hours;
4. Thrombolysis contradictions:

   * Definite cerebral apoplexy history;
   * Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery) or recent trauma to the head or cranium (i.e. < 3 months);
   * Active bleeding or known bleeding disorder/diathesis;
   * Recent administration of any i.v. or s.c. anticoagulation within 12 hours including unfractionated heparin, enoxaparin and/or bivalirudin or current use of oral anticoagulation(warfarin or coumadin);
   * Uncontrolled hypertension, defined as a single blood pressure measurement ≥ 180/110 mm Hg (systolic BP ≥ 180 mm Hg and/or diastolic BP ≥ 110 mm Hg) prior to randomisation;
   * Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current myocardial infarction); Prolonged or traumatic cardiopulmonary resuscitation (> 10 minutes) within the past 2 Weeks Major surgery pending in the following 30 days;
5. Severe complication

   * Other diseases with life expectancy ≤12 months;
   * Any history of Severe renal or hepatic dysfunction(hepatic failure, cirrhosis, portal hypertension and active hepatitis); Neutropenia, thrombocytopenia ; Known acute pancreatitis;
   * Known acute pericarditis and/or subacute bacterial endocarditis;
   * Arterial aneurysm, arterial/venous malformation and aorta dissection;
6. Complex heart condition

   * Cardiogenic shock(SBP <90 mmHg after fluid infusion or SBP<100 mmHg after vasoactive drugs);
   * PCI within previous 1 month or Previous coronary-artery bypass surgery(CABG);
   * Previously known multivessel coronary artery disease not suitable for revascularization;
   * Hospitalisation for cardiac reason within past 48 hours;
7. Not suitable for clinical trial

   * Inclusion in another clinical trial;
   * Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 7 days;
   * Pregnancy or lactating;
   * Body weight <40kg or >125kg;
   * Known hypersensitivity to any drug that may appear in the study;
   * Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
Complete Epicardial and myocardial reperfusion; | Immediately after PCI
  defined as TIMI Flow Grade 3 (TFG 3) for epicardial reperfusion and TIMI Myocardial Perfusion Grade 3 (TMPG 3) for myocardial reperfusionand resolution of the initial sum of ST-segment elevation ≥ 70% in 60 min post catheterisation

SECONDARY OUTCOMES:
TIMI Flow Grade (TFG) | Immediately after PCI
  TIMI Flow Grade (TFG) assesses flow in the epicardial arteries.
TIMI Myocardial Perfusion Grade (TMPG) | Immediately after PCI
  TMPG is an angiographic measure of myocardial perfusion.
ST-segment Resolution | Immediately after PCI
  Resolution of the initial sum of ST-segment elevation ≥ 70%.
TIMI Frame Count (CTFC) | Immediately after PCI
  CTFC is a continuous measurement assessing flow in the epicardial arteries.
TIMI Myocardial Perfusion Frame Count (TMPFC) | Immediately after PCI
  TMPFC is a novel method to standardize and quantify myocardial perfusion by timing the filling and washout of contrast in the myocardium using cine-angiographic frame-counting. Briefly, the first frame of TMPFC was defined as the frame that clearly demonstrated the first appearance of myocardial blush beyond the IRA (F1). The last frame of TMPFC was then defined as the frame where contrast or myocardial blush disappeared (F2). TMPFC is F2-F1 frame counts at a filming rate of 15 frames/sec, or (F2-F1)×2 frame counts at the corrected filming rate of 30 frames/sec.
Wall motion score index (WMSI) by echocardiography | in-hospital and 30 day
  The WMSI will be calculated as the sum of the scores in each segment divided by 16. Each segment will be given a score based on its systolic function (normal = 1, hypokinesis = 2, akinesis = 3).
Clinical Outcomes | 30 days after randomization
  All cause death, non-fatal reinfarction, heart failure, and stroke after randomization constitute the clinical endpoints.

OTHER OUTCOMES:
Main Safety Endpoints-Bleeding events | 30 days after randomization
  Incidence of bleeding events, classified by the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries (GUSTO) severity criteria
Left Ventricular Function | in-hospital and 30 day
  Left ventricular function assessment by echocardiography and cardiac magnetic resonance

CONTACTS AND LOCATIONS:
Overall Officials: Ben He, MD, Study Director — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Canadian Cardiovascular Society; American Academy of Family Physicians; American College of Cardiology; American Heart Association; Antman EM, Hand M, Armstrong PW, Bates ER, Green LA, Halasyamani LK, Hochman JS, Krumholz HM, Lamas GA, Mullany CJ, Pearle DL, Sloan MA, Smith SC Jr, Anbe DT, Kushner FG, Ornato JP, Pearle DL, Sloan MA, Jacobs AK, Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA 2004 guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):210-47. doi: 10.1016/j.jacc.2007.10.001. No abstract available. PMID 18191746
- [Background] Gibson CM. Primary angioplasty compared with thrombolysis: new issues in the era of glycoprotein IIb/IIIa inhibition and intracoronary stenting. Ann Intern Med. 1999 May 18;130(10):841-7. doi: 10.7326/0003-4819-130-10-199905180-00019. PMID 10366375
- [Background] Borgia F, Goodman SG, Halvorsen S, Cantor WJ, Piscione F, Le May MR, Fernandez-Aviles F, Sanchez PL, Dimopoulos K, Scheller B, Armstrong PW, Di Mario C. Early routine percutaneous coronary intervention after fibrinolysis vs. standard therapy in ST-segment elevation myocardial infarction: a meta-analysis. Eur Heart J. 2010 Sep;31(17):2156-69. doi: 10.1093/eurheartj/ehq204. Epub 2010 Jul 2. PMID 20601393
- [Background] Van de Werf F, Bax J, Betriu A, Blomstrom-Lundqvist C, Crea F, Falk V, Filippatos G, Fox K, Huber K, Kastrati A, Rosengren A, Steg PG, Tubaro M, Verheugt F, Weidinger F, Weis M; ESC Committee for Practice Guidelines (CPG). Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J. 2008 Dec;29(23):2909-45. doi: 10.1093/eurheartj/ehn416. Epub 2008 Nov 12. No abstract available. PMID 19004841
- [Background] Ding S, Pu J, Qiao ZQ, Shan P, Song W, Du Y, Shen JY, Jin SX, Sun Y, Shen L, Lim YL, He B. TIMI myocardial perfusion frame count: a new method to assess myocardial perfusion and its predictive value for short-term prognosis. Catheter Cardiovasc Interv. 2010 Apr 1;75(5):722-32. doi: 10.1002/ccd.22298. PMID 19960517
- [Background] Fernandez-Aviles F, Alonso JJ, Pena G, Blanco J, Alonso-Briales J, Lopez-Mesa J, Fernandez-Vazquez F, Moreu J, Hernandez RA, Castro-Beiras A, Gabriel R, Gibson CM, Sanchez PL; GRACIA-2 (Groupo de Analisis de Cardiopatia Isquemica Aguda) Investigators. Primary angioplasty vs. early routine post-fibrinolysis angioplasty for acute myocardial infarction with ST-segment elevation: the GRACIA-2 non-inferiority, randomized, controlled trial. Eur Heart J. 2007 Apr;28(8):949-60. doi: 10.1093/eurheartj/ehl461. Epub 2007 Jan 23. PMID 17244641
- [Derived] Pu J, Ding S, Ge H, Han Y, Guo J, Lin R, Su X, Zhang H, Chen L, He B; EARLY-MYO Investigators. Efficacy and Safety of a Pharmaco-Invasive Strategy With Half-Dose Alteplase Versus Primary Angioplasty in ST-Segment-Elevation Myocardial Infarction: EARLY-MYO Trial (Early Routine Catheterization After Alteplase Fibrinolysis Versus Primary PCI in Acute ST-Segment-Elevation Myocardial Infarction). Circulation. 2017 Oct 17;136(16):1462-1473. doi: 10.1161/CIRCULATIONAHA.117.030582. Epub 2017 Aug 27. PMID 28844990